CLINICAL TRIAL: NCT04405622
Title: Toripalimab Combined With Gemcitabine in Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Toripalimab and Gemcitabine in Recurrent or Metastatic Nasopharyngeal Carcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Chief physician, Proffessor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2020-2104
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Nasopharyngeal Carcinoma; Recurrent Nasopharyngeal Carcinoma; Metastatic Nasopharyngeal Carcinoma; Chemotherapy Effect; Immunotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab plus gemcitabin arm (Experimental): Subjects receive gemcitabine and toripalimab.
  Interventions: Drug: Toripalimab plus gemcitabine

INTERVENTIONS:
Drug: Toripalimab plus gemcitabine — Subjects receive gemcitabine 1000mg/m2 (Day 1 and Day 8) and Toripalimab , 240mg, (Day 1) of each 21 days for at most 6 cycles, followed by Toripalimab 240mg every three weeks (Q3W) maintenance. Treatment was continued until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, or investigator decision.

SUMMARY:
This is an open-label, single center, pilot trial to evaluate the safety and efficacy of toripalimab and gemcitabine in patients with recurrent or metastatic nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; 18-70 years of age.
2. Subjects diagnosed with pathological confirmed metastatic nasopharyngeal carcinoma, or subjects with recurrent NPC that is unfit for local treatment.
3. did't receive any systemic chemotherapy for recurrent and metastatic lesions.
4. Intolerance to or rejection of platinum-based chemotherapy
5. ECOG performance status of 0 or 1.
6. Life expectancy more than 12 weeks.
7. Subjects enrolled must have measurable lesion(s) according to response evaluation criteria in solid (RECIST) v1.1.
8. Adequate organ function assessed by laboratory parameters during the screening period
9. Female subjects agree not to be pregnant or lactating from beginning of the study screening through at least 3 months after receiving the last dose of study treatment. Both men and women of reproductive potential must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy. A highly effective method of contraception is defined as one that results in a low failure rate, that is, less than 1% per year when used consistently and correctly
10. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Subjects with any active autoimmune disease or history of autoimmune disease, or history of syndrome that requires systemic steroids or immunosuppressive medications, including but not limited to the following: rheumatoid arthritis, pneumonitis, colitis (inflammatory bowel disease), hepatitis, hypophysitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Subjects with the following conditions will not be excluded from this study: asthma that requires intermittent use of bronchodilators, hypothyroidism stable on hormone replacement, vitiligo, Graves' disease, or Hashimoto's disease. Additional exceptions may be made with medical monitor approval;
2. Known history of hypersensitivity to any components of the Toripalimab formulation;
3. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration. Note: corticosteroids used for the purpose of IV contrast allergy prophylaxis are allowed;
4. Active central nervous system (CNS) metastases (indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive disease);
5. Uncontrolled clinically significant medical condition, including but not limited to the following:

   1. congestive heart failure (New York Health Authority Class > 2),
   2. unstable angina,
   3. myocardial infarction within the past 12 months,
   4. clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention;
6. Active infection or an unexplained fever; 38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, subjects with tumor fever may be enrolled);
7. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease;
8. Any other medical (eg, pulmonary, metabolic, congenital, endocrinal, or CNS disease), psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results; Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or risk of reactivation based on institutional guidelines and tests. Testing may include the following: HBV DNA, HCV RNA, hepatitis B surface antigen, or anti-Hepatitis B core antibody.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 year
  The safety will be assessed according to CTCAE (V5.0)

SECONDARY OUTCOMES:
The proportion of patients who achieved an objective response | 1 year
  Defined as those with radiologically confirmed complete or partial response according to RECIST 1.1 assessed by the investigator;
The proportion of patients who achieved disease control | 1 year
  Defined as those with RECIST-defined objective response or stable disease according to RECIST 1.1 assessed by the investigator;
The proportion of patients who achieved clinical benefit | 1 year
  Defined as those with confirmed objective response or stable disease that lasted for at least 6 months;
Progression-free survival | 1 year
  Defined from the enrolment to RECIST defined progression or death from any causes;
Duration of response | 1 year
  Defined as the time from first documentation of objective response to radiological disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Ming-Yuan Chen, Guangzhou, Guangdong, China